CLINICAL TRIAL: NCT04220567
Title: Is a Combined Programme of Exercise and Patient-centred Education More Effective Than Exercise Alone in Individuals With Fibromyalgia? A Randomised Controlled Trial
Brief Title: Effectiveness of Exercise and Patient-centred Education on Fibromyalgia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto Politécnico de Setúbal. Escola Superior de Saúde. (Other)
Collaborators: Universidade de Lisboa - Faculdade Letras (Unknown); Centro Hospitalar de Setúbal E.P.E. (Unknown); Centro Hospitalar Lisboa Ocidental (Other Government); Myos - Associação Nacional Contra a Fibromialgia e Síndrome de Fadiga Crónica (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IPSetubalESS_SHARE
Record Dates: First submitted 2020-01-05; First posted 2020-01-07 (Actual); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: Fibromyalgia
Keywords: Fibromyalgia; Exercise; Patient-centred Education; Randomised Controlled Trial
MeSH Terms: conditions — Fibromyalgia; Motor Activity

STUDY DESIGN:
Intervention Model Description: Parallel assignment
Who Masked: Participant, Outcomes Assessor
Masking Description: Double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise and Patient-centred education (Experimental)
  Interventions: Other: Experimental: Exercise and Patient-centred education
- Exercise (Active Comparator)
  Interventions: Other: Active Comparator: Exercise

INTERVENTIONS:
Other: Experimental: Exercise and Patient-centred education — An eight-week programme based on 24 sessions of exercise supervised by a physiotherapist. Exercise will be carried out three times a week. Once a week the exercise session is performed autonomously by patient at home (according to the physiotherapist's recommendations).
  Patient-centred Education will follow the principles of transformative learning & incorporate patients' narratives. It will precede 9 of the 24 exercise sessions and be delivered by the same physiotherapist
  Arms: Exercise and Patient-centred education
Other: Active Comparator: Exercise — An eight-week programme based on 24 sessions of exercise supervised by a physiotherapist. Exercise will be carried out three times a week. Once a week the exercise session is performed autonomously by patient at home (according to the physiotherapist's recommendations).
  Arms: Exercise

SUMMARY:
This study aims to compare the effects of an eight-week exercise and patient-centred education programme with eight-week exercise alone programme on disability, pain intensity, health-related quality of life and patient global impression of change.

A prospective, parallel, double-blinded and multi-centre randomised controlled trial will be carried out.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of fibromyalgia according to the American College of Rheumatology criteria (2016)

Exclusion Criteria:

* Presence of uncontrolled medical disorders (cardiovascular/ metabolic/ neurological/ renal)
* Presence of active oncological disease (or until 5 years and undergoing treatment)
* Presence of inflammatory rheumatic diseases other than fibromyalgia
* Presence of inflammatory osteoarticular disease or severe osteoarthritis (grade IV de Kellgren - Lawrence Classification of Osteoarthritis)
* Previous orthopaedic (column or lower limb) or cardiothoracic surgery in the year before;
* Disability not compatible with the exercise practice required
* Pregnancy
* Attendance to a physiotherapy programme including exercise in the previous three months
* Difficulty in written communication that prevent the fulfilment of self-reported questionnaires.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-01-07 (Actual); Primary Completion 2020-10 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | Baseline
  Measured using the Numeric Pain Rating Scale, NPS, 0-10
Pain intensity | 4 weeks
  Measured using the Numeric Pain Rating Scale, NPS, 0-10
Pain intensity | 8 weeks
  Measured using the Numeric Pain Rating Scale, NPS, 0-10
Pain intensity | Follow-up 3 months
  Measured using the Numeric Pain Rating Scale, NPS, 0-10
Disability and Impact of Fibromyalgia | Baseline
  Measured using the Revised Fibromyalgia Impact Questionnaire, FIQr, 0-100
Disability and Impact of Fibromyalgia | 4 weeks
  Measured using the Revised Fibromyalgia Impact Questionnaire, FIQr, 0-100
Disability and Impact of Fibromyalgia | 8 weeks
  Measured using the Revised Fibromyalgia Impact Questionnaire, FIQr, 0-100
Disability and Impact of Fibromyalgia | Follow-up 3 months
  Measured using the Revised Fibromyalgia Impact Questionnaire, FIQr, 0-100

SECONDARY OUTCOMES:
Neuropathic components in pain | Baseline
  Measured using the painDETECT Questionnaire
Health-related Quality of Life | Baseline
  Measured using the EuroQol 5D 3L, EQ 5D-3L
Health-related Quality of Life | 4 weeks
  Measured using the EuroQol 5D 3L, EQ 5D-3L
Health-related Quality of Life | 8 weeks
  Measured using the EuroQol 5D 3L, EQ 5D-3L
Health-related Quality of Life | Follow-up 3 months
  Measured using the EuroQol 5D 3L, EQ 5D-3L
Patients' perception of improvement or decline in clinical status | 4 weeks
  Measured using the The Patient Global Impression of Change Scale, PGIC, 1-7
Patients' perception of improvement or decline in clinical status | 8 weeks
  Measured using the Patient Global Impression of Change Scale, PGIC, 1-7
Patients' perception of improvement or decline in clinical status | Follow-up 3 months
  Measured using the Patient Global Impression of Change Scale, PGIC, 1-7

CONTACTS AND LOCATIONS:
Locations (1):
- Carmen Caeiro, Setúbal, Portugal